CLINICAL TRIAL: NCT07398807
Title: EFFECTIVENESS OF COMBINING MICRO NEEDLING WITH 5 FLUOROURACIL VERSUS POTENT TOPICAL STEROIDS; IN TREATING LIMITED VITILIGO-RANDOMIZED CONTROLLED STUDY
Brief Title: Effectiveness of Micro-needling With 5 Fluorouracil Versus Potent Topical Steroids in the Treatment of Limited Vitiligo
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital (CMH) institute of Medical Sciences Bahawalpur Pakistan (Other)
Responsible Party: Principal Investigator, Sara Khan, Post graduate resident of Dermatology, Combined Military Hospital (CMH) institute of Medical Sciences Bahawalpur Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1516/EC/14/2025
Record Dates: First submitted 2025-11-15; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Vitiligo
Keywords: Vitiligo; Limited; Microneedling; 5-FU
MeSH Terms: conditions — Vitiligo | interventions — Percutaneous Collagen Induction; Fluorouracil; Clobetasol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Microneedling with topical 5-fluorouracil (Experimental)
  Interventions: Drug: Microneedling with 5-fluorouracil
- Clobetasol propionate 0.05% (Active Comparator)
  Interventions: Drug: Topical application of 0.05% Clobetasol propionate

INTERVENTIONS:
Drug: Microneedling with 5-fluorouracil — Micro-needling will be done, 2 passes will be made on the affected patch of vitiligo with 5 FU. Not more than 0.5 ml 5FU will be used during each session. Session will be repeated 2 weekly for 6 months.
  Arms: Microneedling with topical 5-fluorouracil
Drug: Topical application of 0.05% Clobetasol propionate — Topical 0.05% clobetasol propionate ointment will be applied twice a day on the vitiligo patches.1 finger-tip unit (FTU) will be used for 2% BSA i.e., 0.5 grams.
  Arms: Clobetasol propionate 0.05%

SUMMARY:
The goal of this clinical trial is to learn how well 5 fluorouracil (5FU) with micro-needling works to treat limited vitiligo as compared to strong steroid applied on skin. It will also learn about the safety of both these treatments. The main questions it aims to answer are:

* How well does 5FU with microneedling work to treat vitiligo by returning pigmentation in vitiligo patches as compared to steroid?
* What is participant's satisfaction when treated with 5FU with microneedling as compared to steroid?
* What skin problems do participants have when treated with FU with microneedling and steroid?

Researchers will compare 5FU with microneedling to steroid application to see how well both work to return pigment in vitiligo patches.

Participants will be divided into two groups. For Group A, 5 FU will be rubbed and absorbed on the vitiligo patch after micro-needling every 2 weeks.

For group B, topical 0.05% clobetasol propionate ointment will be applied twice a day on the vitiligo patches for 12 weeks.

Vitiligo patches will be assessed at the start of trial and then after 12 weeks of treatment.

DETAILED DESCRIPTION:
The rationale of this study is to find a cost-effective treatment regime of 5 fluorouracil for limited stable vitiligo. We aim to compare how effective is the combination of micro-needling with 5 Fluorouracil versus topical potent steroids in the cases of stable, limited vitiligo (< 10% body surface area -BSA).

40 patients with limited vitiligo consulting the dermatologist in the hospital OPD will be included in the trial after application of the mentioned inclusion and exclusion criteria. After informed consent, a dermatologist will explain the required details of the procedure to the patients and give them their required treatment plan. They will be randomized into two groups by lottery method.

Demographic data like age, gender, location and number of vitiligo patches will be recorded along with baseline photograph and measurement of the vitiligo patches by VASI score.

In first group i.e., Group A, a topical eutectic mixture of local anesthetic in cream formulation (EMLA) will be applied over the patient's lesions for 30- 45 minutes. Lesion will be cleaned by pyodine iodine applied for at least 5 minutes. Micro-needling will be done by dr. Pen Ultima A6 with 42 needle cartridges (single usage) with 3mm depth and 2 passes will be made on the effected patch of vitiligo. Sterile gauze will be pressed on the lesion for 2 minutes to stop bleeding. Afterwards depth will be decreased to 1.5mm and 5 FU will be rubbed on the lesion before this step. Aim would be to facilitate percutaneous absorption of the drug with micro-needling. Micro-needling device will be held at 90-degree angle and will be glided up and down, followed by side to side and then diagonal sections with light pressure to avoid dragging. Few drops of 5 FU will be rubbed and absorbed again on the vitiligo patch after micro-needling. Not more than 0.5 ml 5FU will be used during each session. Lesions will be covered by a sterile dressing after the procedure. It will be removed after 12 hours. Patient will be instructed to avoid bathing for 24 hours after the procedure. 6 sessions will be done at 2 weeks interval.

Group B will be advised topical 0.05% clobetasol propionate ointment twice a day on the vitiligo patches.1 finger-tip unit (FTU) will be used for 2% BSA i.e., 0.5 grams. The application should be continued for 12 weeks.

A blinded independent medical observer will perform clinical assessment at the end of 12 weeks treatment period using the VASI score and using the following grading scale for all 40 patients: 1, < 25% minimal regain of pigment in the lesion; 2, 26-50% mild regain of pigment in the lesion; 3, 51-75% moderate regain of pigment in the lesion; 4, >75% excellent regain of pigment in the lesion.

Patient satisfaction will also be assessed by grading scale i.e., 1. Not satisfied, 2. Satisfied but partially, 3. Completely satisfied with the treatment.

Side-effects like koebnerization, irritant contact dermatitis, folliculitis and cutaneous atrophy will be noted in both the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study
* Patients of age group of 05 -70 years.
* Vitiligo involving less than or equal to 10% body surface area.

Exclusion Criteria:

* Patients using or have used other treatments for vitiligo
* Pregnant women or lactating women
* Patients with unstable vitiligo
* Patients on immunosuppressant medications due to other diseases
* Patients having anemia, immunosuppression, bleeding disorder, taking anticoagulants or anti-platelet drugs or having epilepsy
* Patient having history of keloids or hypertrophic scars
* Patients with history of hypersensitivity to either of the drugs

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Re-pigmentation of vitiligo patches of patients treated with 5FU with micro-needling versus potent topical steroids at week 12 as assessed by improvement in VASI scores | From enrollment to the end of treatment at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Bahawalpur, Chak Four Hundred Fifty-four, Pakistan